CLINICAL TRIAL: NCT06923553
Title: NDBI Training and Coaching
Brief Title: Implementation of Naturalistic Developmental Behavioral Intervention (NDBI) Through Coaching Caregivers of Young Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, James D Lee, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007006
Record Dates: First submitted 2025-03-27; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Implementation Research
Keywords: Hybrid type 1; autism; NDBI; family coaching; underserved families
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NDBI group (Experimental)
  Interventions: Behavioral: NDBIs

INTERVENTIONS:
Behavioral: NDBIs — Caregivers will meet with clinicians virtually weekly to (a) watch the newly developed NDBI videos that demonstrate the strategy use, (b) discuss how this might be applied to their own child, (c) receive individualized homework planning, (d) record and upload videos of their practice of strategy use with their own child, and (e) review the videos with clinicians to receive individualized feedback on their strategy use. This will occur for 10 weeks. Each session will be video recorded to assess the clinicians' intervention fidelity. After 10 weeks, pre-post tests will be conducted to assess parents' confidence on implementing these strategies, their child's social communication, and satisfaction of providers and caregivers.

SUMMARY:
Naturalistic developmental behavioral interventions (NDBIs) are a newer class of evidence-based interventions for young autistic children to promote their positive developmental or behavioral outcomes. These are often delivered by family members or other natural change agents given the emphasis on naturalistic transactions between an adult and a child. Despite the emerging evidence, there are practical difficulties that hinder wider dissemination and implementation of NDBIs, including low level of access to some of these branded, packaged NDBIs. To mitigate these difficulties related to access, we have created a series of video modules that demonstrate nine commonly used core components in NDBI strategies. In this study, caregivers will receive training and coaching using these modules and both synchronous and asynchronous coaching from a clinician. In this type 1 hybrid implementation trial, there are two groups of participants: (1) caregivers of young autistic children or children with other developmental disabilities/delays, (2) children, and (3) clinicians. Caregivers will meet with clinicians virtually weekly to (a) watch the newly developed NDBI videos that demonstrate the strategy use, (b) discuss how this might be applied to their own child, (c) receive individualized homework planning, (d) record and upload videos of their practice of strategy use with their own child, and (e) review the videos with clinicians to receive individualized feedback on their strategy use. This will occur for 10 weeks. Each session will be video recorded to assess the clinicians' intervention fidelity. After 10 weeks, pre-post tests will be conducted to assess parents' confidence on implementing these strategies, their child's social communication, and satisfaction of providers and caregivers. Qualitative data will also be collected via interviews with some selected participants to gain a deeper understanding of their perceptions.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of a caregiver-mediated intervention incorporating newly developed Naturalistic Developmental Behavioral Intervention (NDBI) modules and clinician coaching. The study consists of: (1) participant recruitment, (2) caregiver training, (3) clinician coaching, (4) data collection, and (5) participant feedback. Below is a detailed description of each phase of the study procedures.

1. Recruitment and Consent Process Recruitment will take place across the United States and Korea, utilizing social media platforms (e.g., Facebook groups), community organizations, and professional networks. Flyers containing a QR code will direct potential participants to a Qualtrics page hosted by UT Austin, where they will receive detailed study information and complete an initial eligibility screening.

   Interested participants will review an embedded informed consent form, which includes a description of study procedures, potential risks, and confidentiality measures. Participants will have the opportunity to ask questions before providing consent. Once consent is obtained, they will complete baseline assessments to collect demographic information and initial measures related to intervention outcomes.
2. Intervention Procedures The intervention consists of 10 weekly sessions (30 minutes each) where trained Board Certified Behavior Analysts (BCBAs) will provide coaching to caregivers on how to implement NDBI strategies in daily interactions with their child. Each session will focus on practicing and refining specific behavioral techniques to promote communication and engagement. Coaching sessions will be conducted via video conferencing (e.g., Zoom) or in-person, depending on participant location.

   Caregivers will receive access to pre-recorded intervention videos demonstrating NDBI techniques, which they are expected to watch before each session. Each video is about 2-3 minutes long and available upon request. The modules are ready for caregivers' viewing online, and it includes topics such as following the child's lead, prompting, prompt fading, natural reinforcement, reciprocal interactions, turn taking, etc.

   To evaluate caregiver strategy implementation, parents will record interactions with their child using a smartphone, tablet, or computer. These interactions will be pre-planned during their weekly session with the clinician who will help plan the specific context, routines, and activities in which the caregivers will practice implementing the strategies that they learned about. Then, caregivers will receive feedback in the next session based on the recordings. These recordings will not exceed 5 minutes in length. The participants will be instructed to only include consented parent and child to ensure privacy of surrounding individuals, if any. These recordings will be uploaded to a secure research platform (e.g., encrypted cloud storage or Qualtrics) for analysis. Videos will be reviewed by research team members to assess strategy fidelity and caregiver engagement.
3. Clinician Coaching and Supervision BCBAs conducting caregiver training will also receive coaching sessions to ensure fidelity in delivering the intervention. These sessions will focus on reviewing caregiver progress, discussing implementation challenges, and refining coaching techniques.

   All clinician coaching sessions will be recorded using Zoom (or another HIPAA-compliant video conferencing platform) and stored on encrypted servers for analysis. These recordings will be used to assess clinician fidelity using a validated fidelity checklist.
4. Data Collection and Outcome Measures

   Participants will complete assessments at baseline (pre-intervention) and post-intervention to measure caregiver skill acquisition, child developmental progress, and intervention effectiveness. The following research measures will be used:
   * Vineland-3 Adaptive Behavior Scale: Assesses child adaptive behavior.
   * WHOQOL (World Health Organization Quality of Life Questionnaire): Measures caregiver well-being.
   * Autism-Specific Parenting Self-Efficacy Scale: Evaluates caregiver confidence in managing their child's behavior.
   * Social Validity Measures (AIM, IAM, FIM): Evaluate caregiver satisfaction and acceptability of the intervention.

   All measures will be administered via Qualtrics to maximize accessibility for participants.
5. Interviews and Focus Group Sessions After completing the intervention, caregivers will participate in structured interviews or focus group discussions to provide qualitative feedback on their experiences. These sessions will be conducted via Zoom or another secure video conferencing platform.

   Participants will have the option to turn off their cameras during discussions to maintain privacy. Interviews and focus groups will be recorded and stored on encrypted servers, with transcripts de-identified before analysis.
6. Data Security and Confidentiality All research activities will take place online to maximize participation and accessibility. Data will be securely stored on password-protected servers, and only authorized research personnel will have access. Video recordings and consent forms will be stored separately from research data, and all identifying information will be de-identified prior to analysis. Additionally, this is a collaborative study that involves UT Austin researchers working with external researchers who are responsible for data collection, analysis of de-identified data, and dissemination of research findings.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers: Primary caregivers of young children aged 0-5 who meet one of the following conditions: (1) diagnosed with autism spectrum disorder, (2) diagnosed with developmental delay, and (3) diagnosed with a developmental disability. Eligible caregivers include: (1) parents, (2) grandparents, (3) legal guardians. All caregivers must be at least 18 years old and must be of Korean descent.
2. Clinicians: The clinicians must hold a current Board Certified Behavior Analyst (BCBA) certification and must have experience delivering behavioral intervention and caregiver training for children aged 0-5.
3. Children: Children in this study must be between 0-5 years old and must have a formal medical diagnosis confirming one of the following conditions: (1) autism spectrum disorder (ASD), (2) developmental delay, or (3) developmental disability.

Exclusion Criteria:

1. Caregivers: Caregivers will be excluded if they (1) primarily care for children over the age of 6, (2) are not Korean speakers, or (3) are unable to fully participate in study activities, such as watching training videos, recording parent-child interactions, or completing required questionnaires.
2. Clinicians: Clinicians will be excluded if they (1) do not hold a valid Board Certified Behavior Analyst (BCBA) certification, (2) lack experience in providing behavioral intervention and caregiver training for children aged 0-5, or (3) only work with children over the age of 6.
3. Children: Children will be excluded if they (1) are older than 5 years, (2) do not have a formal medical diagnosis confirming autism spectrum disorder, developmental delay, or developmental disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vineland-3 Adaptive Behavior Scale | From baseline to the end of treatment at 10 weeks
  The Vineland-3 Adaptive Behavior Composite (ABC) standard score, which summarizes adaptive behavior across domains, has a minimum score of 20 and a maximum score of 160. The higher scores indicate a better outcome.
WHOQOL (World Health Organization Quality of Life Questionnaire) | From baseline to the end of treatment at 10 weeks
  Measures caregiver well-being
Autism-Specific Parenting Self-Efficacy Scale | From baseline to the end of treatment at 10 weeks
  Evaluates caregiver confidence in managing their child's behavior
Acceptability of Intervention Measure | From baseline to the end of treatment at 10 weeks
  4-item instrument measuring caregiver satisfaction and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No